CLINICAL TRIAL: NCT04840810
Title: To Compare the In-plane and Out of Plane Ultrasound Guided Approach for Internal Jugular Vein Cannulation in the Patients Undergoing Elective Cardiac Surgery. A Prospective Randomize Control Trial.
Brief Title: To Compare the In-plane and Out of Plane Ultrasound Guided Approach for Internal Jugular Vein Cannulation in the Patients Undergoing Elective Cardiac Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, Rizwana Shehzad, Staff Medical officer AKUH, Aga Khan University Hospital, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: AgaKhanUH
Record Dates: First submitted 2021-04-08; First posted 2021-04-12 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Catheterization, Central Venous; Ultrasonography; Cardiac Surgical Procedures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Out of plane/ short axis central venous cannulation (Active Comparator): In a short-axis view, the image plane is perpendicular to the course of the vessel and to the needle (needle is "out of plane"). The vessel appears as an anechoic circle on the screen of ultrasound with the needle visualized as a hyperechoic point in cross-section. The central venous cannulation was done in out of plane axis.
  Interventions: Procedure: In-plane Axis
- In-plane/long axis central venous cannulation (Active Comparator): In a long-axis view, the image plane is parallel to the course of the vessel (needle is "in-plane"). The image shows the course of the vessel across the screen and the shaft and point of the needle as it is advanced. The central venous cannulation was done in in-plane axis.
  Interventions: Procedure: Out of plane Axis

INTERVENTIONS:
Procedure: In-plane Axis — In a long-axis view, the image plane is parallel to the course of the vessel (needle is "in-plane"). The image shows the course of the vessel across the screen and the shaft and point of the needle as it is advanced. The central venous cannulation was done in in-plane axis.
  Arms: Out of plane/ short axis central venous cannulation
Procedure: Out of plane Axis — In a short-axis view, the image plane is perpendicular to the course of the vessel and to the needle (needle is "out of plane"). The vessel appears as an anechoic circle on the screen of ultrasound with the needle visualized as a hyperechoic point in cross-section. The central venous cannulation was done in out of plane axis.
  Arms: In-plane/long axis central venous cannulation

SUMMARY:
The insertion of central venous catheters (CVCs) has become an integral part of management of a critically ill patient. Access to the central vein may be required for the administration of hyper osmotic or vasoactive compounds, parenteral nutrition, and rapid infusion of large volumes of fluid or for the continuous or intermittent monitoring of biochemical or physiological parameters. Central venous catheter insertion is also indicated when the insertion of a peripheral line is not possible. Traditionally, CVC insertions have been performed using the landmark technique.

Considering the number of CVCs being inserted every day, this can amount to a large number of complications. Efforts to minimize and prevent the occurrence of complications should be a routine component of quality improvement programs. There is an increasing body of evidence supporting the use of ultrasound guidance for CVC placement.

This makes the strong rationale to conduct this research thus the aim of this study is to evaluate the real benefits i.e outcome of Long versus Short Axis ultrasound guided approach for internal jugular vein cannulation in the patient for elective cardiac surgery as central venous cannulation (CVC).

DETAILED DESCRIPTION:
OBJECTIVE: To compare the in plane and out of plane ultrasound guided approach for internal jugular vein cannulation in the patients undergoing elective cardiac surgery.

Ultrasound-guided central vein cannulation has many advantages, giving the operator the possibility of choosing the most appropriate and safest venous access on the basis of ultrasound assessment, performing a 100% safe insertion, ruling out malposition or pleuropulmonary damages, during and after the procedure.

There is an increasing body of evidence supporting the use of ultrasound guidance for CVC placement.

This makes the strong rationale to conduct this research thus the aim of this study is to evaluate the real benefits i.e outcome of Long versus Short Axis ultrasound guided approach for internal jugular vein cannulation in the patient for elective cardiac surgery as central venous cannulation (CVC).

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted for elective cardiac surgery.
* Age between 18 - 75 years.

Exclusion Criteria:

* BMI more than 30.
* Haemodynamically unstable.
* Patient with abnormal coagulation profile(INR>1.5 or Platelet counts<50,000).
* Patient with a short neck.
* Patient with carotid Atherosclerosis proven on ultrasound.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-04-02 (Actual)

PRIMARY OUTCOMES:
First pass success Rate | immediately after end of procedure
  Recoded in percentage. Needle successfully inserted into the internal jugular vein and there is no need of Readjustment
Duration of procedure | Intraoperative (after skin prick to ultrasound confirmation of presence of guide wire within internal jugular vein)
  Recorded in seconds

SECONDARY OUTCOMES:
Unintentional carotid puncture | immediately after completion of procedure
  Recorded in percentage

CONTACTS AND LOCATIONS:
Locations (1):
- Aga khan university Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schummer W, Schummer C, Rose N, Niesen WD, Sakka SG. Mechanical complications and malpositions of central venous cannulations by experienced operators. A prospective study of 1794 catheterizations in critically ill patients. Intensive Care Med. 2007 Jun;33(6):1055-9. doi: 10.1007/s00134-007-0560-z. Epub 2007 Mar 7. PMID 17342519
- [Background] Jefferson P, Ogbue MN, Hamilton KE, Ball DR. A survey of the use of portable ultrasound for central vein cannulation on critical care units in the UK. Anaesthesia. 2002 Apr;57(4):365-8. doi: 10.1046/j.1365-2044.2002.02319.x. PMID 11939995
- [Background] Randolph AG, Cook DJ, Gonzales CA, Pribble CG. Ultrasound guidance for placement of central venous catheters: a meta-analysis of the literature. Crit Care Med. 1996 Dec;24(12):2053-8. doi: 10.1097/00003246-199612000-00020. PMID 8968276